CLINICAL TRIAL: NCT06694142
Title: Not Always ROSY-Feasibility of Addressing Sexual Dysfunction in Women with Breast and Gynecologic Cancers with a Novel Mobile Application
Brief Title: Feasibility of Addressing Sexual Dysfunction in Women with Breast and Gynecologic Cancers with a Novel Mobile Application
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lavanya Palavalli Parsons, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-24-0817
Record Dates: First submitted 2024-11-07; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Sexual Dysfunction
Keywords: breast and gynecologic cancer patients
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rosy app (Experimental)
  Interventions: Behavioral: Rosy app

INTERVENTIONS:
Behavioral: Rosy app — Participants will be provided a six-month membership subscription to the mobile application ROSY. ROSY will recommend pathways for addressing issues through 1) coaching by board certified coaches or 2) joining a completely anonymous community with other people where they can share experiences and get help as new members of the community to overcome sexual health challenges .Users will work towards their health goals each day using tools from medical and mental health experts . Tools used include 1) virtual workshops and 2) coaching sessions which will provide the opportunity to a) Have an authentic and relatable conversation with an expert b) Explore new pathways to better health experience c) Improve their relationship with themselves, partner, and healthcare providers d) Learn fun ways to improve their everyday wellness e) Access live events from anywhere.

SUMMARY:
The purpose of this study is to identify breast and gynecologic cancer patients with sexual dysfunction, to measure sexual dysfunction with the Female Sexual Function Index (FSFI) and to provide Patients with the opportunity during this six-month period to follow up with a healthcare provider to discuss the sexual dysfunction needs and to see if a medical intervention can be of aid.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a current or historic diagnosis of breast cancer or gynecologic cancer (uterine ovarian, fallopian tube, peritoneal, cervical, vulva, or vaginal cancers)
* Agree to participate in the study with completion of survey and use of ROSY mobile application

Exclusion Criteria:

* Currently pregnant
* Non-English speaking (ROSY is currently is only available is in English).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-11-18 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Change in sex related personal distress as assessed by the Female Sexual Function Index (FSFI) | Baseline, 6 months
  FSFI is a 19-item instrument that measures 6 domains of sexual function: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. This uses a Likert-type scale, with scores ranging from 0 to 5, except for questions 1, 2, 13, and 16, which are scored from 1 to 5. The total score ranges from 2.0 to 36.0, with higher scores indicating better functioning.
Change in sexual dysfunction as assessed by the Social Determinants of Health (SDOH) questionnaire | Baseline, 6 months
  score ranges from 0 to 10, higher score showing worse outcome

SECONDARY OUTCOMES:
Change in sex related personal distress as assessed by the Female Sexual Function Index (FSFI) in ethnic minority groups | end of study (6 months after baseline)
  FSFI is a 19-item instrument that measures 6 domains of sexual function: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. This uses a Likert-type scale, with scores ranging from 0 to 5, except for questions 1, 2, 13, and 16, which are scored from 1 to 5. The total score ranges from 2.0 to 36.0, with higher scores indicating better functioning.
Change in sex related personal distress as assessed by the Female Sexual Function Index (FSFI) in sexual and gender minority groups | end of study (6 months after baseline)
  FSFI is a 19-item instrument that measures 6 domains of sexual function: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. This uses a Likert-type scale, with scores ranging from 0 to 5, except for questions 1, 2, 13, and 16, which are scored from 1 to 5. The total score ranges from 2.0 to 36.0, with higher scores indicating better functioning.
Change in sex related personal distress as assessed by the Female Sexual Function Index (FSFI) in unpartnered women | end of study (6 months after baseline)
  FSFI is a 19-item instrument that measures 6 domains of sexual function: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. This uses a Likert-type scale, with scores ranging from 0 to 5, except for questions 1, 2, 13, and 16, which are scored from 1 to 5. The total score ranges from 2.0 to 36.0, with higher scores indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Lavanya P Parsons, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No